CLINICAL TRIAL: NCT05813886
Title: Evaluation of Dynamic Balance After Recovery From COVID 19 Disease
Status: Completed | Type: Observational
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Amira Mohamed Afify, Associate professor, October 6 University
Other Study IDs: P.T.REC/012/003590
Record Dates: First submitted 2023-04-11; First posted 2023-04-14 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 Respiratory Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: biodex balance system — The balance tests of the patients were performed 2 to24 WEEKS after their recovery from the disease, which was confirmed by the evaluations of the Covid-19 staff and negative polymerase chain reaction test.

SUMMARY:
effect of post covid-19 on dynamic balance in patients after recovery from covid-19 disease.

DETAILED DESCRIPTION:
effect of post covid-19 on dynamic balance in patients after recovery from COVID disease.

patients will treated with medical protocol of COVID 19 an out-patient clinic , and followed up by the chest specialist . The balance tests of the patients were performed 2 to 14 weeks after their recovery from the disease, which was confirmed by the evaluations of the COVID staff and negative polymerase chain reaction test.the patients will evaluated using questionnaires. First, the question will whether feeling in balance in the daily life or not. The answer will classified as "yes"or "no". Second, asked to fill "Dizziness Handicap Inventory"(DHI), which is a multidimensional self- assessment scale created to evaluate the effects of dizziness and balance problems on the quality of life as well as the level of disability of the patients. Assess balance , which consists of a movable balance platform that provides up to 20 of surface tilt in a 360 range of motion. The platform is interfaced with computer software that enables the device to serve as an objective assessment of balance . The measure of postural stability includes the overall (OA), the anteroposterior (AP) and the mediolateral (ML) stability scores. A high score in the OA index indicates poor balance. The OA stability score is believed to be the best indicator of the overall ability of the patient to balance the platform

ELIGIBILITY:
Inclusion Criteria:

* 25post COVID-19 patients suffering from inbalance.
* Age will be ranged from 30 to 40 years old.
* Body mass index (BMI) will be ranged from 25 to 35 Kg/m2.
* Diagnosed as COVID-19 patients with a positive reverse transcription polymerase chain reaction (RT-PCR) result of SARS-CoV-2, or typical computerized tomography (CT) evidence of viral pneumonia.
* All enrolled patients with moderate covid-19 infection.

Exclusion Criteria:

* Severe disease or hospitalization at intensive care units will excluded from the study.
* Patients with previous hearing problems or balance disorders.
* Patients who had ear surgery, cardiovascular and circulatory problems,.
* Patients with orthopedic problems in the lower extremities due to other problems
* Patients with Any history of neurological or psychiatric disease, severe visual or auditory impairments.
* Diabetic patients.

Ages: 30 Years to 40 Years | Sex: All
Age Groups: Adult
Gender Based: Yes — MALE AND FEMALE
Study Population: 25 patients (males and females) who recovered from Covid-19 disease will be selected from 6 october unversity Hospital outpatient Clinic their age from 30 -40 years old and 25 healthyage and gender matched (males and females
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
overall (OA), the anteroposterior (AP) and the Medio lateral (ML) stability scores | 2 to24 WEEKS after their recovery from the disease
  A high score in the OA index indicates poor balance. The OA stability score is believed to be the best indicator of the overall ability of the patient to balance the platform

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 u, El-Sheikh Zayed City, Giza Governorate, Egypt